CLINICAL TRIAL: NCT05863013
Title: Longitudinal Changes in the ADL-Glittre Test in Patients With Lung Cancer: Pre- and Postoperative Analysis Using Rehabilitation in a Randomized Controlled Trial
Brief Title: Use of the ADL-Glittre Test in the Pre and Postoperative Period of Patients With Lung Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67676823.4.0000.5259
Record Dates: First submitted 2023-03-25; First posted 2023-05-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer, Nonsmall Cell; Quality of Life; Physical Disability; Surgery
Keywords: ADL-Glittre test; Functional capacity; pulmonary rehabilitation; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients included in the study will be evaluated:
  T0 (baseline): Baseline assessments will be performed immediately prior to randomization and will include lung function [spirometry, measurement of pulmonary CO2 diffusing capacity (DLCO) and measurement of respiratory muscle strength], handgrip measurement , measurement of quadriceps strength (HR ), exercise capacity (TGlittre1), level of physical activity in daily life (International Physical Activity Questionnaire - IPAQ) and assessment of QoL (St. George's Respiratory Questionnaire - SGRQ).
  T1 (day before surgery): Patients will repeat lung function, HGS measurement, HR measurement, TGlittre2, IPAQ, and SGRQ.
  T2 (1 month after surgery): Patients will repeat the tests from the previous phase.
  Data on postoperative complications and 30-day complications and mortality will also be recorded.
  T3 (4 months after surgery): Patients will have repeat lung function, HGS measurement, HR measurement, TGlittre4, IPAQ, and SGRQ.
Who Masked: Outcomes Assessor
Masking Description: The sample will be divided into two groups: Intervention Group and Control Group. Patients meeting the inclusion criteria will be randomly assigned to one of 2 groups (GI and CG) in a 1:1 ratio using a computer-generated random allocation sequence using the stratified block randomization method of SAS version 9.1. 3 (SAS Institute, Cary, NC, USA). Randomization will be performed by an independent research assistant who will not participate in any other phase of this study. The health professionals who will work in the study (physicians and physiotherapists) will be informed of the assignment of the treatment by telephone confirmation. The evaluators of clinical and statistical results will be "blinded" to the randomization, since it was not feasible to "blind" the other professionals involved in the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health education and home care (No Intervention): They will receive standard care: a therapeutic education session on admission, plus daily in-house early postoperative rehabilitation, delivered by a physiotherapist. The therapeutic educational session will involve counseling and self-care management, aiming to prepare patients for the postoperative period, emphasizing breathing exercises and sputum clearance techniques, pain control strategies and self-care. It will consist of smoking cessation education, respiratory retraining (pursed-lip breathing, diaphragmatic breathing, and segmental breathing), and secretion clearance training (coughing exercise, huffing, assisted coughing, and postural drainage).
- Pulmonary rehabilitation (Experimental): They will receive standard care described (AP) plus perioperative PR, with 20 preoperative and 60 postoperative sessions. The preoperative sessions will be held 2X/week, in addition to the home sessions 3X/week. Each outpatient session will last 2 hours and will consist of therapeutic education, aerobic exercises, resistance training of lower limbs, upper limbs and abdominal wall, and respiratory muscle training (RMT), which will include breathing pattern, positive expiratory pressure and inspiratory muscles training and home will last for 1h, unsupervised and personalized MRT plus 30 min of aerobic walking at an intensity of 60-80% of maximum HR. Participants will receive a portable pedometer and HR monitor. Postoperative rehabilitation will be offered only to the IG, from 1 month after surgery, with 60 sessions divided into 24 outpatient sessions performed 2X/week and 36 home sessions 3X/week. The postoperative program will last 12 weeks.
  Interventions: Other: ADL-Glittre Test

INTERVENTIONS:
Other: ADL-Glittre Test — They will receive standard care described plus perioperative pulmonary rehabilitation, with 20 preoperative sessions and 60 postoperative sessions. Preoperative sessions will be held 2X/week, in addition to home sessions 3X/week. Each outpatient session will last 2 hours and will consist of therapeutic education, aerobic exercises, resistance training of lower limbs, upper limbs and abdominal wall and respiratory muscle training (RMT), which will include breathing pattern, positive expiratory pressure and training of inspiratory and respiratory muscles. home will last 1h, unsupervised and personalized MRT plus 30 min of aerobic walking at 60-80% of maximum HR intensity. Participants will receive a portable pedometer and HR monitor. Postoperative rehabilitation will be offered only to the IG, from 1 month after surgery, with 60 sessions divided into 24 outpatient sessions performed 2X/week and 36 home sessions 3X/week. The postoperative program will last 12 weeks.
  Arms: Pulmonary rehabilitation

SUMMARY:
Lung cancer is the most common type of cancer and the leading cause of cancer death worldwide, in both men and women. Improvements in earlier preoperative staging and more effective adjuvant treatment have improved survival in non-small cell lung cancer, although surgical resection remains the mainstay of care for all patients in stages I to IV.

This study proposes to evaluate the functional capacity through TGlittre in patients with non-small cell lung cancer, before and after thoracic surgery, taking into account the predictive role of this test in the risk of complications and in the evaluation of the impact of functional rehabilitation.

DETAILED DESCRIPTION:
In the population of patients with lung cancer, two critical points that constitute gaps in the literature are: 1) the definition of operability using only pulmonary function tests and the consequent preparation of the patient for the surgical act; and 2) the postoperative approach and the consequent screening aimed at improving quality of life and reducing morbidity. In addition to the sophistication of pulmonary rehabilitation that has occurred in recent decades, the ADL-Glittre test was also developed, which is a measure of submaximal effort that assesses functional capacity and encompasses several tasks that simulate activities of daily living involving both lower limbs the higher, being an easy to administer, valid and reliable test to measure the functional status. This study proposes to evaluate the functional capacity through TGlittre in patients with non-small cell lung cancer, before and after thoracic surgery, taking into account the predictive role of this test in the risk of complications and in the evaluation of the impact of functional rehabilitation. As specific objectives, this study seeks to: test the reliability and validity of TGlittre in patients with non-small cell lung cancer; compare the results of TGlittre with those of lung function and quality of life in the pre- and postoperative period; to determine the impact of the preoperative pulmonary rehabilitation program on performance on the TGlittre; to determine the impact of the postoperative PR program on TGlittre performance; and to evaluate the incidence of postoperative complications and length of stay, considering the performance in TGlittre and the performance in the PR program. Using block randomization, participants who meet the inclusion criteria will be randomly assigned to one of 2 groups: 1) Intervention Group: Pulmonary Rehabilitation; and 2) Control Group: Standard Care. PR will be performed pre- and postoperatively, lasting 4 and 12 weeks, respectively. These participants will submit to the following tests: International Physical Activity Questionnaire; St. George's Respiratory Questionnaire; lung function (spirometry, measurement of lung diffusion capacity to carbon monoxide and measurement of respiratory muscle strength); handgrip strength; quadriceps strength; and TGlittre. The aim of this study is to support the applicability of TGlittre as an evaluative strategy for pulmonary rehabilitation in the pre- and postoperative periods of patients with non-small cell lung cancer, and also to verify the impact of pre- and postoperative rehabilitation strategies on quality of life, morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSCLC stages I to IV, that is, those patients without evidence of mediastinal disease or local organ invasion.
* Age equal to or greater than 18 years.
* The following types of lung surgery: pneumonectomy, bilobectomy, lobectomy, segmentectomy and wedge resection.
* Resection by thoracotomy or video-assisted thoracoscopic surgery.

Exclusion Criteria:

* Patients known to need adjuvant treatments.
* Show inability to walk.
* Not being able to perform pulmonary function tests and/or functional tests.
* Presence of cardiovascular, neurological or orthopedic diseases.
* Bronchopleural fistula, sudden increase in chest drainage or active intrathoracic hemorrhage, chylothorax or other serious adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Functional capacity through the Glittre Activities of Daily Living test (ADL-Glittre test). | six months
  The participant must complete 5 laps in the shortest possible time. The test consists of carrying a backpack containing a 2.5kg weight completing a circuit with the following activities. The participant rises from a seated position and walks on a 10-m flat course, interposed halfway by a stairway with 2 steps to ascend and 2 to descend. After completing the course, the individual approaches a 2-teir shelf containing 3 objects weighing 1kg each, placed on the highest shelf (shoulder height), that must be moved 1 by 1 to the bottom shelf (waist height) and then down to the floor. Then, the objects are placed on the bottom shelf again and finally on the top shelf. Then, the individual turns and walks back over the course; immediately after completion of 1 lap, another lap is started, completing the same circuit. The instructions are standardized, and there is no incentive during the test. Two tests are performed with a minim.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | six months
  The International Physical Activity Questionnaire (IPAQ) contains seven open questions and aims to quantify the weekly time spent in physical activities of moderate and vigorous intensity, in different everyday contexts, such as work, transportation, household chores and leisure, and also the time spent in passive activities performed in a sitting position. To answer the questions, participants will be instructed to consider the week before the IPAQ application date and will subsequently be classified according to the level of activity as sedentary, irregularly active, active or very active, according to the weekly frequency and duration of activities performed.
St. George's Respiratory Questionnaire (SGRQ) | six months
  To measure quality of life, the Saint George Hospital questionnaire on respiratory disease was applied, which was validated and adapted for the Brazilian population. This instrument covers aspects in three domains, which are: symptoms, activity and psychosocial impacts that the disease can influence in their daily routine. The answers translate into points that, once added together, can infer about an altered Quality of life in a given domain. A score is calculated for each domain (0-100 points) and a total score is also calculated, the higher the score, the worse the measured quality of life.
Handgrip strength (HGS) | six months
  HGS will be measured in kilograms using a handheld digital dynamometer (SH5001, Saehan Corporation, Korea). The HGS will be evaluated with the participants sitting in a chair without arms, with elbow flexion at 90°, forearms in a neutral position and extension wrist angle between 0 and 30°. The maximum force will be evaluated after sustained contraction of 3s in the dominant hand; the highest value of 3 attempts with 1 min intervals will be considered for analysis.
Quadriceps strength | six months
  Quadriceps strength will be assessed using a traction dynamometer with a sensor capacity of 200 kg (E-lastic 5.0, E-sport SE, Brazil). The amplitude of movement in the execution of the test will be determined in 90°, starting from 90° with the knee in flexion. Maximum strength will be evaluated after a sustained contraction of 5 s on the dominant leg, and the highest value from 3 attempts with 1-min intervals will be considered for analysis.
Spirometry- forced expiratory volume in one second (FEV1) | six months
  During the spirometry test, the individual must remain seated, with the head in a neutral position to avoid changes in expiratory flows. The evaluator must advise that the maneuvers are performed through encouragement and verbal stimulation. The procedure must be guided and demonstrated by the technician, through a tube. It is necessary for the patient to perform a maximum inspiration, followed by a rapid and sustained expiration. The measure of forced expiratory volume in one second (FEV1) will be evaluated, which is the amount of air eliminated in the first second of the forced expiratory maneuver.
Spirometry- Forced Vital Capacity (FVC) | six months
  During the spirometry test, the measurement of forced vital capacity (FVC) will also be evaluated, which can be identified through the volume eliminated in the forced expiratory maneuver from total lung capacity to residual volume.
Spirometry- Peak Expiratory Flow (PEF) | six months
  During the spirometry test, the peak expiratory flow (PEF) will also be evaluated, which represents the maximum air flow during the FVC maneuver. PEF is an effort-dependent expiratory parameter that reflects the caliber of the proximal airways and is often used as an effective cough marker.
Carbon monoxide diffusion capacity (DLCO) | Six months
  For the DLCO analysis, the use of a nose clip will be requested (in order to avoid nasal breathing), remaining in a sitting position and coupling to the pulmonary function device through an appropriate mouthpiece. After slow expiration to residual volume, rapid but not forced inspiration will be performed. Upon reaching full lung capacity, an inspiratory pause of approximately 10s will occur and then the inhaled gas will be exhaled smoothly and without interruptions. The expired air volume will be collected for analysis that will determine the difference between inspired CO and expired CO (diffused CO).
Respiratory muscle strength | Six months
  For analysis of respiratory muscle strength, measurements of inspiratory pressure and maximum expiratory pressure will be recorded. The individual must remain in a sitting position, with the head in a neutral position and is asked to perform a maximum expiration, that is, up to the residual volume, to measure the inspiratory pressure. Next, the patient makes a maximal inspiratory effort against the occluded airway. To verify the expiratory pressure, the patient is instructed to perform a maximum inspiration up to the level of total lung capacity, then, they must perform a maximum expiratory effort against the occluded airway. The maximum value of three maneuvers that varied less than 20%, the variability within the measurements, the predicted value, and the lower limit of normality range will be recorded. National equations will be adopted to calculate the predicted values of each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almquist D, Khanal N, Smith L, Ganti AK. Preoperative Pulmonary Function Tests (PFTs) and Outcomes from Resected Early Stage Non-small Cell Lung Cancer (NSCLC). Anticancer Res. 2018 May;38(5):2903-2907. doi: 10.21873/anticanres.12537. PMID 29715115
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] de Araujo CL, Karloh M, Dos Reis CM, Palu M, Mayer AF. Pursed-lips breathing reduces dynamic hyperinflation induced by activities of daily living test in patients with chronic obstructive pulmonary disease: A randomized cross-over study. J Rehabil Med. 2015 Nov;47(10):957-62. doi: 10.2340/16501977-2008. PMID 26538411
- [Background] Araujo LH, Baldotto C, Castro G Jr, Katz A, Ferreira CG, Mathias C, Mascarenhas E, Lopes GL, Carvalho H, Tabacof J, Martinez-Mesa J, Viana LS, Cruz MS, Zukin M, Marchi P, Terra RM, Ribeiro RA, Lima VCC, Werutsky G, Barrios CH; Grupo Brasileiro de Oncologia Toracica. Lung cancer in Brazil. J Bras Pneumol. 2018 Jan-Feb;44(1):55-64. doi: 10.1590/S1806-37562017000000135. PMID 29538545
- [Background] Arikan H, Yatar I, Calik-Kutukcu E, Aribas Z, Saglam M, Vardar-Yagli N, Savci S, Inal-Ince D, Ozcelik U, Kiper N. A comparison of respiratory and peripheral muscle strength, functional exercise capacity, activities of daily living and physical fitness in patients with cystic fibrosis and healthy subjects. Res Dev Disabil. 2015 Oct-Nov;45-46:147-56. doi: 10.1016/j.ridd.2015.07.020. Epub 2015 Aug 1. PMID 26241869
- [Background] Assis ACB, Lopes AJ. Functional exercise capacity in rheumatoid arthritis unrelated to lung injury: A comparison of women with and without rheumatoid disease. J Back Musculoskelet Rehabil. 2022;35(2):449-458. doi: 10.3233/BMR-210056. PMID 34275888
- [Background] Boujibar F, Gillibert A, Gravier FE, Gillot T, Bonnevie T, Cuvelier A, Baste JM. Performance at stair-climbing test is associated with postoperative complications after lung resection: a systematic review and meta-analysis. Thorax. 2020 Sep;75(9):791-797. doi: 10.1136/thoraxjnl-2019-214019. Epub 2020 Jul 10. PMID 32651199
- [Background] Bradley A, Marshall A, Stonehewer L, Reaper L, Parker K, Bevan-Smith E, Jordan C, Gillies J, Agostini P, Bishay E, Kalkat M, Steyn R, Rajesh P, Dunn J, Naidu B. Pulmonary rehabilitation programme for patients undergoing curative lung cancer surgery. Eur J Cardiothorac Surg. 2013 Oct;44(4):e266-71. doi: 10.1093/ejcts/ezt381. Epub 2013 Aug 19. PMID 23959742
- [Background] Bray F, Laversanne M, Weiderpass E, Soerjomataram I. The ever-increasing importance of cancer as a leading cause of premature death worldwide. Cancer. 2021 Aug 15;127(16):3029-3030. doi: 10.1002/cncr.33587. Epub 2021 Jun 4. PMID 34086348
- [Background] British Thoracic Society; Society of Cardiothoracic Surgeons of Great Britain and Ireland Working Party. BTS guidelines: guidelines on the selection of patients with lung cancer for surgery. Thorax. 2001 Feb;56(2):89-108. doi: 10.1136/thorax.56.2.89. No abstract available. PMID 11209097
- [Background] Brunelli A, Xiume F, Refai M, Salati M, Marasco R, Sciarra V, Sabbatini A. Evaluation of expiratory volume, diffusion capacity, and exercise tolerance following major lung resection: a prospective follow-up analysis. Chest. 2007 Jan;131(1):141-7. doi: 10.1378/chest.06-1345. PMID 17218568
- [Background] Brunelli A, Salati M. Preoperative evaluation of lung cancer: predicting the impact of surgery on physiology and quality of life. Curr Opin Pulm Med. 2008 Jul;14(4):275-81. doi: 10.1097/MCP.0b013e328300caac. PMID 18520258
- [Background] Brunelli A, Kim AW, Berger KI, Addrizzo-Harris DJ. Physiologic evaluation of the patient with lung cancer being considered for resectional surgery: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e166S-e190S. doi: 10.1378/chest.12-2395. PMID 23649437
- [Background] Bui KL, Nyberg A, Maltais F, Saey D. Functional Tests in Chronic Obstructive Pulmonary Disease, Part 2: Measurement Properties. Ann Am Thorac Soc. 2017 May;14(5):785-794. doi: 10.1513/AnnalsATS.201609-734AS. PMID 28244801
- [Background] Cavalheri V, Donaria L, Ferreira T, Finatti M, Camillo CA, Cipulo Ramos EM, Pitta F. Energy expenditure during daily activities as measured by two motion sensors in patients with COPD. Respir Med. 2011 Jun;105(6):922-9. doi: 10.1016/j.rmed.2011.01.004. Epub 2011 Jan 28. PMID 21276720
- [Background] Cesario A, Ferri L, Galetta D, Pasqua F, Bonassi S, Clini E, Biscione G, Cardaci V, di Toro S, Zarzana A, Margaritora S, Piraino A, Russo P, Sterzi S, Granone P. Post-operative respiratory rehabilitation after lung resection for non-small cell lung cancer. Lung Cancer. 2007 Aug;57(2):175-80. doi: 10.1016/j.lungcan.2007.02.017. Epub 2007 Apr 17. PMID 17442449
- [Background] Choi J, Yang Z, Lee J, Lee JH, Kim HK, Yong HS, Lee SY. Usefulness of Pulmonary Rehabilitation in Non-Small Cell Lung Cancer Patients Based on Pulmonary Function Tests and Muscle Analysis Using Computed Tomography Images. Cancer Res Treat. 2022 Jul;54(3):793-802. doi: 10.4143/crt.2021.769. Epub 2021 Oct 20. PMID 34696566
- [Background] Colice GL, Shafazand S, Griffin JP, Keenan R, Bolliger CT; American College of Chest Physicians. Physiologic evaluation of the patient with lung cancer being considered for resectional surgery: ACCP evidenced-based clinical practice guidelines (2nd edition). Chest. 2007 Sep;132(3 Suppl):161S-77S. doi: 10.1378/chest.07-1359. PMID 17873167
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] de Alegria SG, Kasuki L, Gadelha M, Lopes AJ. The Glittre Activities of Daily Living Test in patients with acromegaly: Associations with hand function and health-related quality of life. J Back Musculoskelet Rehabil. 2021;34(3):441-451. doi: 10.3233/BMR-200089. PMID 33492273
- [Background] de Groot PM, Wu CC, Carter BW, Munden RF. The epidemiology of lung cancer. Transl Lung Cancer Res. 2018 Jun;7(3):220-233. doi: 10.21037/tlcr.2018.05.06. PMID 30050761
- [Background] de Oliveira Vacchi C, Martha BA, Macagnan FE. Effect of inspiratory muscle training associated or not to physical rehabilitation in preoperative anatomic pulmonary resection: a systematic review and meta-analysis. Support Care Cancer. 2022 Feb;30(2):1079-1092. doi: 10.1007/s00520-021-06467-4. Epub 2021 Aug 21. PMID 34417883
- [Background] Fugazzaro S, Costi S, Mainini C, Kopliku B, Rapicetta C, Piro R, Bardelli R, Rebelo PFS, Galeone C, Sgarbi G, Lococo F, Paci M, Ricchetti T, Cavuto S, Merlo DF, Tenconi S. PUREAIR protocol: randomized controlled trial of intensive pulmonary rehabilitation versus standard care in patients undergoing surgical resection for lung cancer. BMC Cancer. 2017 Jul 31;17(1):508. doi: 10.1186/s12885-017-3479-y. PMID 28760151
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] Goldsmith I, Chesterfield-Thomas G, Toghill H. Pre-treatment optimization with pulmonary rehabilitation in lung cancer: Making the inoperable patients operable. EClinicalMedicine. 2020 Nov 30;31:100663. doi: 10.1016/j.eclinm.2020.100663. eCollection 2021 Jan. PMID 33554075
- [Background] Graham BL, Brusasco V, Burgos F, Cooper BG, Jensen R, Kendrick A, MacIntyre NR, Thompson BR, Wanger J. 2017 ERS/ATS standards for single-breath carbon monoxide uptake in the lung. Eur Respir J. 2017 Jan 3;49(1):1600016. doi: 10.1183/13993003.00016-2016. Print 2017 Jan. PMID 28049168
- [Background] Hirpara DH, Kidane B, Rogalla P, Cypel M, de Perrot M, Keshavjee S, Pierre A, Waddell T, Yasufuku K, Darling GE. Frailty assessment prior to thoracic surgery for lung or esophageal cancer: a feasibility study. Support Care Cancer. 2019 Apr;27(4):1535-1540. doi: 10.1007/s00520-018-4547-9. Epub 2018 Nov 14. PMID 30426204